CLINICAL TRIAL: NCT05882513
Title: A Prospective, Single-arm, Single-center, Exploratory Study of the Safety and Efficacy of Serplulimab Combined With Chemotherapy in Patients With Resectable Non-small-cell Lung Cancer
Brief Title: Serplulimab Combined With Chemotherapy in Patients With Resectable Non-small-cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0485
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: NSCLC; Neoadjuvant Therapy
Keywords: serplulimab; Non small cell lung cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung cancer group (Experimental): Squamous cell carcinoma: Serplulimab: 4.5mg/kg, i.v, day1; albumin paclitaxel 260mg/m2, day1; carboplatin AUC=5, i.v, day1.
  Non-squamous cell carcinoma: Serplulimab: 4.5mg/kg, i.v, day1 ; pemetrexed 500mg/m2, day1 ; carboplatin AUC=5, i.v, day1.
  Preoperative neoadjuvant therapy for 3 cycles, one cycle every 21 days. Surgical resection of lung cancer will be arranged about 4-8 weeks after the last cycle of neoadjuvant therapy.
  Interventions: Drug: Serplulimab and neoadjuvant therapy; Procedure: surgical resection of lung cancer; Other: Tumour will be Collected from participant. Fate of sample is Destruction after use

INTERVENTIONS:
Drug: Serplulimab and neoadjuvant therapy — Squamous cell carcinoma: Serplulimab: 4.5mg/kg, i.v, day1; albumin paclitaxel 260mg/m2, day1; carboplatin AUC=5, i.v, day1.
  Non-squamous cell carcinoma: Serplulimab: 4.5mg/kg, i.v, day1 ; pemetrexed 500mg/m2, day1 ; carboplatin AUC=5, i.v, day1.
  Other Names: Serplulimab
Procedure: surgical resection of lung cancer — radical resection of lung cancer
  Other Names: Surgery
Other: Tumour will be Collected from participant. Fate of sample is Destruction after use — Tumour sample will be collected after surgery

SUMMARY:
China with high incidence of non-small cell lung cancer. In the past few decades, surgery, radiotherapy, chemotherapy and other treatments were continuously improved, however, the mortality of lung cancer patients was not significantly decreased. For patients with locally advanced lung cancer, direct surgery is not effective. It is difficult to achieve radical resection by surgery merely, and even if many patients receive surgery, they may eventually have tumor recurrence and poor survival rate. Therefore, it is necessary to explore effective perioperative neoadjuvant treatment to reduce the risk of postoperative recurrence and improve the postoperative survival rate of patients. According to the reports, PD-1/ PD-L1 immunocheckpoint inhibitor may become a new method for the treatment of lung cancer. Preliminary clinical results showed that immunotherapy combined with chemoradiotherapy provided a synergies antitumor effect. Multiple clinical results showed that serplulimab provided higher overall response rate for advanced lung cancer. However, in patients with locally advanced lung cancer, the efficacy of serplulimab combined with chemotherapy for sequential radical surgery is still unclear. The purpose of this study is to observe and evaluate the efficacy and safety of serplulimab combined with chemotherapy in the neoadjuvant therapy of resectable non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent;
2. patients age 18 to 75 years old
3. primary resectable, histologically confirmed non small cell lung cancer;
4. non small cell lung cancer the clinical stage was IIA-IIIB (no N3 patient) (according to AJCC TNM stage, 8th edition).
5. ECOG PS 0-1.
6. the diseases could be resectable assessed by thoracic oncologist

Exclusion Criteria:

1. with significant cardiovascular disease;
2. current treatment with anti-viral therapy or HBV;
3. Female patients who are pregnant or lactating;
4. history of malignancy within 5 years prior to screening;
5. active or history of autoimmune disease or immune deficiency;
6. signs of distant metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (PCR) | 1 month after surgery
  No residual invasive tumor cells were found in the pathological examination of resected specimens,including the primary tumor and lymph nodes.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | 1 month after surgery
  In the pathological examination of resected specimens, the proportion of residual tumor cells was less than 10%.
Objective Response Rate (ORR) | before surgery
  The proportion of subjects with imaging PR or CR assessed according to RECIST 1.1 criteria
2-year and 5-year overall survival | 2-year and 5-year after enrolled
  The proportion of all study cases in which no death from any cause occurred within 2 years and 5 years after enrolled
Incidence of Treatment-related Adverse Events | 1 month after surgery
  Incidence of Treatment-related Adverse Events as Assessed by CTCAE v5.0
R0 resection rate | 1 month after surgery
  The pathological results will showed that the incision margin was negative and no residual cancer cells were found under the microscope
The changes in the tumor tissue sample among non-PCR (NPCR) and PCR patients | 3 month after surgery
  By using mass spectrometry (CyTOF) and single-cell analysis, we comprehensively characterized the immune landscape in the tumor sample of patients after anti-PD-1 immunotherapy, aiming to explore the immune subsets correlated with neoadjuvant immunotherapy response.

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Wang, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China, China